CLINICAL TRIAL: NCT06836765
Title: Expression of FosB Gene in Laryngeal Cancer Tissues and It's Clinical Prognosis Significance
Brief Title: The Relationship Between the Differential Expression of FosB Protein in Laryngeal Cancer Tissues and Clinical Prognosis
Status: Not yet recruiting | Type: Observational
Sponsor: Yang ji (Other)
Responsible Party: Sponsor-Investigator, Yang ji, associate professor, Neijiang No.2 People's Hospital
Organization: Neijiang No.2 People's Hospital (Other)
Other Study IDs: NeijiangPH2
Record Dates: First submitted 2024-08-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Laryngeal Carcinoma
Keywords: Laryngeal cancer; FosB(FBJ murine osteosarcoma viral oncogene homolog B) gene; Immunohistochemistry; Cox regression analysis
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — the investigators shall are Collecting 100 to 200 cases of laryngeal cancer patients who have been finally diagnosed and treated in our institution. In order to make pathological sections,the investigators will are Collect their laryngeal cancer pathological tissues and adjacent tissues of these paitents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The expression of FosB positive group: Researcher will incorporate the positive expression of FosB protein in laryngeal cancer tissues into the positive study group by immunohistochemical methods!
  Interventions: Other: the expression positive in laryngeal cancer tissue
- The expression of FosB negative group: Researcher will incorporate the positive expression of FOSB protein in laryngeal cancer tissues into the positive study group and vice versa into the negative study group by immunohistochemical methods!
  Interventions: Other: the expression negative in laryngeal cancer tissue

INTERVENTIONS:
Other: the expression negative in laryngeal cancer tissue — Researcher will incorporate the positive expression of FOSB protein in laryngeal cancer tissues into the positive study group and vice versa into the negative study group by immunohistochemical methods!
  Groups: The expression of FosB negative group
Other: the expression positive in laryngeal cancer tissue — Researcher will incorporate the positive expression of FOSB protein in laryngeal cancer tissues into the positive study group and vice versa into the negative study group by immunohistochemical methods!
  Groups: The expression of FosB positive group

SUMMARY:
To determine whether there is statisstical difference in FosB (FBJ murine osteosarcoma viral oncogene homolog B) protein expression between laryngeal cancer tissue and adjacent tissue through immunohistochemistry methods.

If there are differences, further the investigators will collect relevant patients information,such as clinical stages, pathological types, clinical prognosis and so on. ultimately analyze whether it is related to the expression of FOsB in laryngeal cancer tissue and adjacent tissues

DETAILED DESCRIPTION:
First,the investigators will collect 100 to 200 cases of laryngeal cancer patients who have been finally diagnosed and treated in our institution in the past five years. Laryngeal cancer pathological tissues and adjacent tissues will be selected to make pathological sections. Use immunohistochemistry to confirm the differences in FosB protein between laryngeal cancer tissues and adjacent tissues, and clarify whether there are differences.

secondly,if there are differences, further the investigators will collect relevant patients information,such as clinical stages, pathological types, clinical prognosis and so on. Review the clinical data of corresponding patients, including age, gender, smoking and alcohol history, clinical stages, pathological types and clinical prognosis, etc., and compare whether there are statistical differences.

Finally, clinical prognostic data of relevant patients were collected through outpatient follow-up, online and telephone follow-up, to determine whether there is a correlation between Fosb expression in laryngeal cancer tissue and clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

* laryngeal squamous cell carcinoma was diagnosed ,and biopsy was confirmed by two pathologists;
* Primary tumor of Laryngeal ,and there was no distant metastasis;
* Standard treatment such as surgery and Preliminarily-diagnosed parients;
* full clinical and pathological data information and good follow-up;
* there was no previous fatal diseases such as complicated tumors.

Exclusion Criteria:

* Secondary cancer or cancer with distant metastasis;
* Patients who have not seen a doctor for the first time or have received surgery or radiotherapy or chemotherapy in other hospitals;
* Clinical and pathological data were missing and loss to follow-up;
* Patients who abandoned treatment or standard treatment procedures has not been completed;
* The past medical history of other lethal diseases such as complicated tumors.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Researchers are Collecting 100 to 200 cases of laryngeal cancer patients who have been finally diagnosed and treated in research institution.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
the number of fosb gene positive expression cases in laryngeal carcinoma cells and adjacent tissues was determined. | one month
  the number of fosb gene positive expression cases in laryngeal carcinoma cells and adjacent tissues was determined by immunohistochemical test of pathological sections.

SECONDARY OUTCOMES:
_Experimental result of western blot and PCR._Correlation analysis data between clinical information and experimental results.. | three months
  Researcher will verify the effection of FosB gene on the proliferation and migration of Hep-2 laryngeal cancer cells through a series of basic experiments,such as Immunohistochemistry,western blot,PCR,and so on.clinical prognoostic information of patients was collected and the relationship with fosb gene expression was analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Cllinical Laboratory of Chuanbei Medical College, Nanchong, China/SiChuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eferl R, Wagner EF. AP-1: a double-edged sword in tumorigenesis. Nat Rev Cancer. 2003 Nov;3(11):859-68. doi: 10.1038/nrc1209. No abstract available. PMID 14668816
- [Background] Liu S, Luan J, Ding Y. miR-144-3p Targets FosB Proto-oncogene, AP-1 Transcription Factor Subunit (FOSB) to Suppress Proliferation, Migration, and Invasion of PANC-1 Pancreatic Cancer Cells. Oncol Res. 2018 Jun 11;26(5):683-690. doi: 10.3727/096504017X14982585511252. Epub 2017 Jun 24. PMID 28653602
- [Background] Hung YP, Fletcher CD, Hornick JL. FOSB is a Useful Diagnostic Marker for Pseudomyogenic Hemangioendothelioma. Am J Surg Pathol. 2017 May;41(5):596-606. doi: 10.1097/PAS.0000000000000795. PMID 28009608